CLINICAL TRIAL: NCT02135432
Title: A Randomized, Double-Blind, Placebo Controlled Pilot Study to Determine the Safety and Efficacy of Ivacaftor (VX-770) for the Treatment of Chronic Obstructive Pulmonary Disease (The TOPIC Trial)
Brief Title: TOPIC Trial for COPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Steven M Rowe, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F140319002; TOPIC Trial (Other: UAB)
Record Dates: First submitted 2014-04-15; First posted 2014-05-12 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive pulmonary disease, Ivacaftor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivacaftor (VX-770) (Experimental): twice a day administration of Ivacaftor: 150mg
  Interventions: Drug: Ivacaftor
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivacaftor
  Other Names: Kalydeco
  Arms: Ivacaftor (VX-770)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, multiple-dose, pilot study of orally-administered ivacaftor in subjects with chronic obstructive pulmonary disease. Subjects will be administered the study drug ivacaftor 150 mg (or placebo) twice daily (BID).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 40-65
* A clinical diagnosis of COPD as defined by GOLD
* At Least a 10 pack year smoking history
* Exhibit symptoms of chronic bronchitis defined by MRC
* FEV1% predicted ≥ 35% and ≤70% Post Bronchodilator
* Clinically stable in the last 4 weeks with no evidence of COPD exacerbation
* Weight of 40 kg-120 kg
* Willingness to use at least one form of acceptable birth control including abstinence, condom with spermicide, or hormonal contraceptives
* Willing to monitor blood glucose if known history of diabetes mellitus requiring insulin or medical therapy

Exclusion Criteria:

* Current Diagnosis of Asthma
* Daytime use of Oxygen Therapy
* Documented history of drug abuse within the last year
* Subjects should not have a pulmonary exacerbation or changes in therapy for pulmonary disease within 28 days before receiving the first dose of study drug.
* Cirrhosis or elevated liver transaminases > 3X ULN
* GFR < 50 estimated by Cockcroft-Gault
* Any illness of abnormal lab finding that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Pregnant or Breastfeeding
* Subjects taking any inhibitors or inducers of CYP3A4, including certain herbal medications and grapefruit/grapefruit juice.
* Uncontrolled Diabetes
* Excluded medications and foods include the drugs and foods provided in the appendix document.
* Clinically significant arrhythmias or conduction abnormalities that in the opinion of the investigator affect patient safety have been added as exclusion criteria and criteria for withdrawal.

Patients who have not been stable or have been hospitalized in the past 3 months with any clinically significant cardiac conditions.

Subjects with history of cancer (current or past, unless remote (>5years))except for localized non-melanomatous skin cancers History of Stroke/CVA History of myocardial infarction/acute coronary syndrome Cardiac Failure NYHC grade III-IV Diabetes Type I Uncontrolled Hypertension Primary or secondary pulmonary hypertension

-

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivacaftor (VX-770): twice a day administration of Ivacaftor: 150mg
  Ivacaftor
- Placebo: matching placebo
  Placebo
Period: Overall Study
Arm/Group | Ivacaftor (VX-770) | Placebo
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivacaftor (VX-770) | Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Full Range); unit: years] | 55 [49 to 65] | 62 [60 to 65] | 55 [49 to 65]
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 2 | 1 | 3
Gender [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in COPD as Measured by the Sweat Analysis in Each Group
Description: sweat analysis is measured by performing a sweat test in each participant. The primary analysis will compare the within group change in sweat chloride before (day 1) and after (day 14) ivacaftor or placebo administration and will be used to test the null hypothesis of no change in sweat chloride using a paired t-test unless the distributions are notably skewed, in which case the non-parametric Wilcoxon signed-rank test will be implemented due to small sample size.
Time Frame: baseline to 2 weeks
Population: 8 patients were analyzed in the ivacaftor Arm because 8 patients were randomized to study drug and only 4 patients were randomized in the placebo arm because 4 patients received placebl
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ivacaftor (VX-770) | Placebo
Number analyzed (Participants) | 8 | 4
mmol/L | -8.0 (4.4) | 2.0 (1.5)

2. Secondary Outcome: Change in COPD as Measured by Nasal Potential Difference
Description: Evaluate the efficacy of ivacaftor treatment in patients with COPD including measures of CFTR activity and clinical outcome as measured by change in nasal potential difference measurement in each group. These data will be used to test the null hypothesis of no change in nasal potential difference (ΔLow Chloride plus isoproterenol) using a paired t-test unless the distributions are notably skewed, in which case the non-parametric Wilcoxon signed-rank test will be implemented due to small sample size.
Time Frame: baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: millivolts
Groups:
- Ivacaftor: patients randomized to ivacaftor twice daily
Arm/Group | Ivacaftor | Placebo
Number analyzed (Participants) | 8 | 4
millivolts | -4.9 (3.9) | 1.0 (6.4)

3. Secondary Outcome: Number of Adverse Events Experienced by the Ivacaftor Subjects and Placebo Subjects.
Description: Number of adverse events per subject in each the Ivacaftor subjects and placebo subjects
Time Frame: baseline to 2 weeks
Measure: Number; unit: adverse events
Arm/Group | Ivacaftor (VX-770) | Placebo
Number analyzed (Participants) | 8 | 4
adverse events | 22 | 14

4. Secondary Outcome: Change in COPD as Measured by Change in Percentage of FEV1 as Measured in Each Group
Description: Spirometry will be analyzed by ATS criteria, and the best of three reproducible efforts will be used to calculate FEV1 in comparison to Hankinson standards. The primary analysis will be the change in FEV1% from day 0 to day 14 within subject, and will be tested against the null hypothesis that no change occurs using a paired t-test unless the distributions are notably skewed, in which case the non-parametric Wilcoxon signed-rank test will be implemented due to small sample size.
Time Frame: baseline to 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of FEV1
Arm/Group | Ivacaftor (VX-770) | Placebo
Number analyzed (Participants) | 8 | 4
percentage of FEV1 | -2.3 (5.2) | 1.8 (9.3)

5. Other Pre Specified Outcome: Pharmacokinetics as Described by AUC12 of Subjects Receiving Ivacaftor
Time Frame: baseline to 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Ivacaftor (VX-770) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/4
Other Adverse Events (participants affected / at risk) | 7/8 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivacaftor (VX-770) (N=8) | Placebo (N=4)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivacaftor (VX-770) (N=8) | Placebo (N=4)
decreased/diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0)
Loose Stools (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
this pilot trial was under powered and potentially too brief to detect definitive changes in lung function

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No